

| SOCIAL BEHAVIORAL INSTRUCTIONS AND TEMPLATE | | |
|---------------------------------------------|-----------|--------|
| NUMBER | DATE | PAGE |
| HRP-503a | 3/22/2021 | 1 of 8 |

#### Instructions and Notes:

- Depending on the nature of what you are doing, some sections may not be applicable to your research. If so, mark as "NA".
- When you write a protocol, keep an electronic copy. You will need a copy if it is necessary to make changes.

#### 1 Protocol Title

Include the full protocol title: Innovative Family Prevention with Latinos in Disadvantaged Settings

#### 2 Background and Objectives

Provide the scientific or scholarly background for, rationale for, and significance of the research based on the existing literature and how will it add to existing knowledge.

- Describe the purpose of the study.
- Describe any relevant preliminary data or case studies.
- Describe any past studies that are in conjunction to this study.

By 2050, 35% of US children will be Latinos<sup>1</sup>, and these youth will number 28 million in the US public schools. Latino youth are at disproportionate risk for growing up in poverty, attending economically disadvantaged schools, and being exposed to stressors associated with their minority status. Yet, they are under-represented in prevention science. When included in trials, Latinos have low rates of recruitment and retention. Yet evidenced-based family programs designed to enhance protective factors (interpersonal and socio-emotional competencies; positive family dynamics) can buffer the negative impacts of contextual adversity. Thus, identifying efficacious programs that can successfully engage youth and parents in economically disadvantaged settings is critical for Latino youth, for their families, and for the nation. The proposed project tests the efficacy of a family-focused program. This innovative program is focused on sibling relationships and parenting of siblings as synergistic targets of change to promote positive interpersonal family dynamics and parent and youth psychosocial and behavioral health and well-being. This translational effort builds on strong theoretical and empirical premises including a successful pilot study (Updegraff et al., 2017; ASU SIBS Program, IRB ID 1208009477). Using a rigorous design and measurement, aims are to: (a) test the efficacy of SIBS, delivered via 12 weekly afterschool sibling sessions and 3 family nights in the familiar elementary school setting, versus a contact-equivalent attention control condition; and (b) test whether cultural resources (familism values), sociocultural risks, and sibling dyad characteristics (birth order, sibling and sibling dyad gender constellation) moderate program efficacy. Mexican-origin sibling dyads (5th graders and younger siblings; N = 390 dyads) and their parents will be recruited from economically disadvantaged elementary schools and randomly assigned within school to intervention or contact-equivalent attention control conditions. Assessments will be conducted at pre-test, post-test, and 18-month follow-up, and include: (a) interviews/surveys with parents and target siblings; (b) teacher ratings and school grades; and (c) daily diary data collected on 7 consecutive days from each sibling. We will test program effects on short- and long-term outcomes, including siblings' socio-emotional skills and adjustment, school engagement and achievement, daily positive and negative well-being, family relationship quality, and siblings' and parents' global psychosocial well-being. Findings will advance prevention science by identifying an efficacious program that capitalizes on cultural assets to promote positive family dynamics and psychosocial well-being among Latinos, including by incorporating daily measurements of intervention targets and outcomes to identify mechanisms underlying program effects.

#### 3 Data Use

Describe how the data will be used. Examples include:

- Dissertation, Thesis, Undergraduate honors project
- Publication/journal article, conferences/presentations
- Results released to agency or organization
- Results released to participants/parents
- Results released to employer or school
- Other (describe)

The primary purpose of the project will be to disseminate publications and presentations. It is possible that students involved in the project may propose to use data for a dissertation, thesis, or undergraduate honor's project. At the completion of the study, summaries will be sent to the schools that participated in the project.



| SOCIAL BEHAVIORAL INSTRUCTIONS AND TEMPLATE | | |
|---------------------------------------------|-----------|--------|
| NUMBER | DATE | PAGE |
| HRP-503a | 3/22/2021 | 2 of 8 |

#### 4 Inclusion and Exclusion Criteria

Describe the criteria that define who will be included or excluded in your final study sample. If you are conducting data analysis only describe what is included in the dataset you propose to use.

Indicate specifically whether you will target or exclude each of the following special populations:

- Minors (individuals who are under the age of 18)
- Adults who are unable to consent
- Pregnant women
- Prisoners
- Native Americans
- Undocumented individuals

We propose a sample of 390 sibling dyads (i.e., 5th grader and his/her next youngest sibling in the 1st through 4th grade). Parents in these families will be invited to participate; participation of one parent is required, but all parents/guardians living in the home will be invited to participate.

#### 5 Number of Participants

Indicate the total number of participants to be recruited and enrolled: 390 5th graders; 390 younger siblings in the 1st through 4th grade; 390 primary parents; up to 390 second parents as available in each family.

#### 6 Recruitment Methods

- Describe who will be doing the recruitment of participants.
- Describe when, where, and how potential participants will be identified and recruited.
- Describe and attach materials that will be used to recruit participants (attach documents or recruitment script with the application).

Letters will be sent home through the collaborating school districts (see letter of support from Mesa School District). Follow-up phone calls will be made by bilingual project staff who will be hired if the project is funded. We will work with the school districts to identify Latino 5<sup>th</sup> graders and send a introductory letter to each family (sent home via the classroom teachers).

Eligibility includes a 5<sup>th</sup> grader and younger sibling (1st to 4<sup>th</sup> grade) attending the same elementary school and being of Mexican origin, as defined by parents' reports of whether each sibling has a biological parent, grandparent, or earlier ancestor who was of Mexican heritage. Families who meet the study's eligibility criteria and are willing to participate will be scheduled for a home visit. During the home visit conducted by group leaders in both intervention and attention-control conditions (so that they can establish rapport with children and parents toward program involvement and retention), we will introduce families to the project, review the procedures, obtain informed consent (for parents; including consent to contact children's teachers and obtain school grades) and assent (for siblings). We also will schedule daily diary calls with target siblings and the pre-test phone interview (45-60 min) with parents. After pre-test data are collected from parents, youth, and teachers, families will be randomized to control or intervention group within each school.

A modification will be submitted with recruitment letters and screening script if the study is funded. These materials will be submitted in English and Spanish along with a translation certificate. Letters of permission from the collaborating schools will be submitted via modification prior to any work beginning in the schools. We have included the letter of support for the grant from the Mesa School District. We would obtain updated support for this specific project if funded and submit as a modification.

#### 7 Procedures Involved

Describe all research procedures being performed, who will facilitate the procedures, and when they will be performed. Describe procedures including:

- The duration of time participants will spend in each research activity.
- The period or span of time for the collection of data, and any long term follow up.
- Surveys or questionnaires that will be administered (Attach all surveys, interview questions, scripts, data collection forms, and instructions for participants to the online application).
- Interventions and sessions (Attach supplemental materials to the online application).
- Lab procedures and tests and related instructions to participants.
- Video or audio recordings of participants.
- Previously collected data sets that that will be analyzed and identify the data source (Attach data use agreement(s) to the online
  application).



| SOCIAL BEHAVIORAL INSTRUCTIONS AND TEMPLATE | | |
|---------------------------------------------|-----------|--------|
| NUMBER | DATE | PAGE |
| HRP-503a | 3/22/2021 | 3 of 8 |

<u>Data collection.</u> First, data will be collected via phone interviews at all three assessments from one parent or parents depending on who agrees to participate (mothers and fathers living together in the children's primary residence will both be invited). Youth reports will be collected separately with 5<sup>th</sup> graders and younger siblings in afterschool sessions (pre- and post-test), and in a home visit (18-month follow-up given that many children may have changed schools over this period). Afterschool sessions will last a total of 90 minutes, including a bathroom break, snack time, survey administration (about 45 minutes), and a game or activity at the end. Items are read aloud and responses recorded by interviewers for younger children. For 5<sup>th</sup> graders, survey items are read to small groups (3 to 4 children) and each child records his/her responses on a paper survey.

Due to COVID-19, and the closing of AZ K-12 schools (likely for the remainder of the school year), we are requesting a modification to our protocol for youth surveys. Youth surveys were typically administered in the afterschool setting. The procedures (script, survey) will remain the same but we will conduct it over the phone with children (a revised version for this new format is included). Due to the difficulty of mailing the goody bags (and the expense), which is the normal incentive, we request approval to pay each child \$10 for their participation in the survey over the phone. This payment is the equivalent of the costs of the goody bags for children. The money would be added to the checks sent to parents, due to not being able to send cash in the mail and the inability to deliver payments in person due to COVID-19 social distancing restrictions per the CDC. This procedure would be for the remaining post-program surveys from our intervention cohort for this year (Cohort 2), and our one-year follow-up assessment with children in April (Cohort 1 of the study).

Next, 7 "daily diary" calls will be conducted with each sibling on consecutive evenings about an hour before children's bedtimes (adapted from the Daily Inventory of Stressful Experiences-Youth (DISE-Y). These calls (about 15 minutes each) focus on children's experiences with target sibling and parents, their use of intervention skills, and their psychosocial well-being during the call day. The daily diary calls will be conducted by the Penn State Survey Research Center. Survey questions for parents and children and for the daily phone calls are attached to this application.

As part of the informed consent process we will request permission from parents to contact each child's teacher to complete measures of achievement and functioning in the school setting. If parents agree, a letter describing the study and a copy of the questionnaires for that child, identified by ID number, will be sent to the teacher. Each form is underlined.

#### Recruitment:

- 1). Recruitment Letter and Flyer sent home via school;
- 2). Families are contacted using the recruitment screening script.

Home Visit with Each Family (families who are eligible and agree):

Home visit script used to conduct each visit.

- 1). Parent Consent and Child Assent
- 2). <u>Emergency Authorization Form</u> (information needed for group leaders who are conducting intervention sessions with children)



| SOCIAL BEHAVIORAL INSTRUCTIONS AND TEMPLATE | | |
|---------------------------------------------|-----------|--------|
| NUMBER | DATE | PAGE |
| HRP-503a | 3/22/2021 | 4 of 8 |

- 3). <u>Tracer Authorization</u> and <u>Tracer Letters</u> completed by each family so that we do not lose them between assessment points. This is a strategy that is common with low-income, highly mobile samples like ours and used in all of our prior studies at ASU.
- 4). Family Demographics (background characteristics asked of parents during the home visit)
- 5). <u>Payment Form</u> (completed in person so that the checks can be mailed after phone interviews; required by petty cash).

# **Pre-Test Surveys**

- 1). Parent Surveys (with at least one parent, but both when present and consent)
- 2). 5<sup>th</sup> grader survey and younger sibling survey administered to children during afterschool session using the child survey administration protocol.
- 3). <u>Daily Phone Calls</u> administered over the phone to children by the Penn State Survey Research Center using <u>Child Diary C1</u>.
- 3). <u>Teacher Demographics</u> and <u>Teacher Reports of Child Functioning Survey</u> (requested of teachers of participating children if parents provide consent during home visit to contact teachers)
- 4). Nightly Phone Calls conducted by Penn State Survey Research Center

#### Intervention

After pre-test data are collected, families will be randomized to control or intervention group within each school. Both conditions include twelve weekly afterschool sessions (90 minutes each) and three family nights, all conducted in the familiar school setting. For both conditions, incentives for program participation include snacks for sibling sessions and, for family nights, dinner for families, child care for non-target siblings, and money for gas or transportation.

- 1. Intervention Condition: SIBS Manual C1 Final
- 2. Control Condition: Academic Skills Manual C1 Final

### **Family Night Feedback Forms**

<u>Feedback forms</u>: Collected anonymously from parents to get their feedback about the program. The forms are done in English and Spanish and there is one version for the SIBS curriculum (FFN Feedback Form SIBS\_Eng and Spa) and then a version for the control (Academic Skills) curriculum (FFN Feedback Form AS\_Eng and Spa).

#### **Post-Test**

- 1. Parent Post-Test (English and Spanish) titled SIBS\_Parent Post-Test ENG/SPA C1
- 2. Parent Feedback Forms (SIBS curriculum, Academic Skills Curriculum, English and Spanish) titled SIBS Parent AS/SIBS Prog Feedback C1 Eng/Spa.
- 3. Parent Interview English and Spanish (SIBS Parent Post Test C1 Eng and Spa)
- 4. Family Background Questions (English and Spanish in a single document; SIBS Parent\_Post-Test Background C1 Eng Span)



| SOCIAL BEHAVIORAL INSTRUCTIONS AND TEMPLATE | | |
|---------------------------------------------|-----------|--------|
| NUMBER | DATE | PAGE |
| HRP-503a | 3/22/2021 | 5 of 8 |

- 5. 5<sup>th</sup> Grader/Younger Sibling Survey English and Spanish (5<sup>th</sup> Grade/Younger Sibling Post Test C1 Eng and Span
- 6. Teacher Survey
- 7. Parent Survey Administered with <u>Parent Survey Script</u> and child survey administered with <u>Child</u> Post-Test Protocol
- 8. Revised child protocol to administer post-program surveys over the phone.

# **One-Year Follow-Up**

- 1. Script to contact families in English and Spanish (English and Spanish included) ALREADY APPROVED.
- 2. Family Background Parent Survey (English and Spanish)
- 3. Parent Survey (the only new items are Section 2e in Version A and 4e in Version B, and Section 3d "Life Events" in both versions) English and Spanish versions incuded.
- 4. Child Survey (6<sup>th</sup> Grade Survey includes five new items: Section 3, Items 3, 6, 9, 12, and 15. There are no new items in the younger sibling survey). English and Spanish versions included.
- 5. 6<sup>th</sup> Grader Teacher Survey (no new items) English only (no Spanish needed).

#### 8 Compensation or Credit

- Describe the amount and timing of any compensation or credit to participants.
- Identify the source of the funds to compensate participants
- Justify that the amount given to participants is reasonable.
- If participants are receiving course credit for participating in research, alternative assignments need to be put in place to avoid coercion.



| SOCIAL BEHAVIORAL INSTRUCTIONS AND TEMPLATE | | |
|---------------------------------------------|-----------|--------|
| NUMBER | DATE | PAGE |
| HRP-503a | 3/22/2021 | 6 of 8 |

Each family will receive \$35 for participation of the primary parent, \$35 for phone interviews, and \$35 for participation of a 2<sup>nd</sup> parent (if available and agrees) at pre-test. Honorarium at post-test is \$40 for primary parent, phone interviews, and second parent, and \$50 at 18-month follow-up. This will include a home visit to complete initial paperwork and informed consent and assent, interviews with each parent (about 90 minutes each), after school sessions with each child initial home visit and interview (90 minutes), and the 7 nightly diary calls with the siblings (about 2 additional hours across 7 days for each child). Parents also will provide transportation home from school after the afterschool sessions. Thus, the monetary amount recognizes their total investment of time for each wave of data collection. For the intervention sessions (program and control), incentives for program participation include snacks for sibling sessions and, for family nights, dinner for families, child care for non-target siblings, money for gas or transportation, and a raffle for each of the three family nights for a gift card or movie tickets to encourage a family activity. Teachers also complete surveys and receive \$10/survey.

Addition for Cohorts 2 and 3: We have added a \$20 payment for the families' time for the home visit, which requires about an hour for parents and two children. Because this takes up a greater amount of time than in our prior studies and because we do some of the parent background information during this visit, we have added the home visit payment to compensate families for their time. The consent form has been revised.

We are familiar with the ASU policy FIN 421-05 and have followed this policy in our prior longitudinal work. We will confirm that participants are receiving less than \$600 within a calendar year. For those receiving more, we will complete the appropriate tax forms. We will comply with all procedures as outlined in this policy as we have done in the past.

#### 9 Risk to Participants

List the reasonably foreseeable risks, discomforts, or inconveniences related to participation in the research. Consider physical, psychological, social, legal, and economic risks.

The risks of the surveys, interviews, and daily diary phone calls utilized for data collection in this study are very low. Some participants may feel uncomfortable answering questions about personal behavior. Other potential risks include threats to privacy or confidentiality posed by the collection of personal data, including reports of antisocial or illegal behavior.

The risks associated with the intervention and control condition programming are also very low. Family members will be asked to join in group meetings in which discussions, role-plays, and fun activities are employed to teach relationship skills. The risks associated with these activities are equivalent to those in everyday life.

#### 10 Potential Benefits to Participants

Realistically describe the potential benefits that individual participants may experience from taking part in the research. Indicate if there is no direct benefit. Do **not** include benefits to society or others.

While there are no direct benefits to children and families from participation in the data collection, findings to date suggest that intervention group participants may benefit from the activities included in the proposed program. Family relationships may become closer and more cohesive, and both parents and children may experience increases in well-being. Sibling relationship dynamics, in particular, may be enhanced, and youth adjustment outcomes may improve.



| SOCIAL BEHAVIORAL INSTRUCTIONS AND TEMPLATE | | |
|---------------------------------------------|-----------|--------|
| NUMBER | DATE | PAGE |
| HRP-503a | 3/22/2021 | 7 of 8 |

#### 11 Privacy and Confidentiality

Describe the steps that will be taken to protect subjects' privacy interests. "Privacy interest" refers to a person's desire to place limits on with whom they interact or to whom they provide personal information. Click here for additional guidance on <u>ASU Data Storage Guidelines</u>.

Describe the following measures to ensure the confidentiality of data:

- Who will have access to the data?
- Where and how data will be stored (e.g. ASU secure server, ASU cloud storage, filing cabinets, etc.)?
- How long the data will be stored?
- Describe the steps that will be taken to secure the data during storage, use, and transmission. (e.g., training, authorization of access, password protection, encryption, physical controls, certificates of confidentiality, and separation of identifiers and data, etc.).
- If applicable, how will audio or video recordings will be managed and secured. Add the duration of time these recordings will be kept.
- If applicable, how will the consent, assent, and/or parental permission forms be secured. These forms should separate from the rest of the study data. Add the duration of time these forms will be kept.
- If applicable, describe how data will be linked or tracked (e.g. masterlist, contact list, reproducible participant ID, randomized ID, etc.).

If your study has previously collected data sets, describe who will be responsible for data security and monitoring.

To ensure confidentiality, collected data will be de-identified: data collection forms will have numeric IDs. Only the PIs and key research personnel (program coordinator, project directors at ASU and Penn State) will have access to individually identifiable private information about human subjects (e.g., lists matching participants and IDs). This information will be kept electronically on two password-protected servers in password-protected files (secure servers at ASU and Penn State), and a hard copy will be kept in a locked filing cabinet housed within a locked office space (Cowden 137) separate from where the data will be kept (Cowden 207). Consent/assent forms will be kept in Cowden 137 in a locked file cabinet separate from the data. Consent/assent and the master ID list will be destroyed within one year after all data collection is complete; data will be kept until five years after the last publication as specified by the American Psychological Association. As required by ASU, all study personnel (staff, students at both ASU and Penn State) will complete the CITI training when hired for the project.

#### 12 Consent Process

Describe the process and procedures process you will use to obtain consent. Include a description of:

- Who will be responsible for consenting participants?
- Where will the consent process take place?
- How will consent be obtained?
- If participants who do not speak English will be enrolled, describe the process to ensure that the oral and/or written information
  provided to those participants will be in that language. Indicate the language that will be used by those obtaining consent.
   Translated consent forms should be submitted after the English is approved.



| SOCIAL BEHAVIORAL INSTRUCTIONS AND TEMPLATE | | |
|---------------------------------------------|-----------|--------|
| NUMBER | DATE | PAGE |
| HRP-503a | 3/22/2021 | 8 of 8 |

Initial contact regarding participation in the study will be made via letters sent through collaborating elementary schools, with follow-up phone calls (or home visits to families who do not have a phone) to assess parents' interest and eligibility. Parents who agree to be screened for eligibility and those who meet eligibility requirements will be scheduled for a home visit. During home visits, trained bilingual (English and Spanish) project staff will present the informed consent forms to parents and the assent forms to youth (after informed consent is completed by parents). The consent process informs potential participants about the study and explains that participation is voluntary and that participants have the right to discontinue involvement at any time. Risks are enumerated in the informed consent form and described orally during the consent process. Parents will sign consent forms for themselves and give consent on behalf of their participating child. Parents will also be asked to provide consent for researchers to contact teachers and obtain school report card grades. The consent process will take place in person. All recruitment and informed consent materials will be available in both Spanish and English. Participants will be informed of the limits of this confidentiality, which are in cases of suspected child abuse or neglect, and harm to self or others (such as intimate partner or child). Confidentiality regulations and limits to these regulations will be adhered to as follows: The two PIs have expertise in directing and running prevention studies and are mandated reporters required to report child abuse as required by law.

We will conduct interviews with children in a private location in the school/home so that their answers cannot be overheard. Because the diary phone calls require only that children respond yes/no or to a rating scale, concern about privacy/confidentiality is mitigated. Teacher questionnaires will be pre-coded with a family/child ID and data will be returned by mail to the project office in individual, pre-addressed, stamped envelopes, which likewise mean that risk for privacy/confidentiality violations is minimal. Teachers will also be instructed to maintain confidentiality in their responses.

All updated materials will be submitted in Spanish via a modification after the English versions are approved. We do this as follows: Materials are translated from English to Spanish and back translated from Spanish to English after the English versions of study materials are approved. A third individual will then review both versions for equivalency and discrepancies will be resolved by the team. A translation certificate will be submitted after signed by the forward and back translators. This will be completed as a modification to the study. We have followed this protocol in all of our prior work with Mexican-origin families and are familiar with and have substantial expertise in conducting research with English and Spanish-speaking Latino/Mexican-origin families (see (Updegraff et al., 2017; ASU SIBS Program, IRB ID 1208009477).

#### 13 Training

Provide the date(s) the members of the research team have completed the CITI training for human participants. This training must be taken within the last 4 years. Additional information can be found at: Training.

Updegraff (PI) - training is on file with IRB. Completion date was September 23, 2017.

Additional team members can be found in the staff table as a separate document, updated each year with new staff members.

# ASU SIBS Project Arizona State University

# T. Denny Sanford School of Social and Family Dynamics

Informed Consent for Parents/Legal Guardians and Minors

#### INTRODUCTION

The purpose of this form is to provide you (as a prospective research study participant) information that may affect your decision as to whether or not to participate in this research and to record the consent of those who agree to be involved in the study.

### **RESEARCHER**

Dr. Kimberly Updegraff, a professor of Family and Human Development at Arizona State University, has invited you to participate in a research study.

#### **DESCRIPTION OF RESEARCH STUDY**

The purpose of this research study is to evaluate the effectiveness of a program to promote positive sibling and family relationships, peer relationships, and school adjustment. If you decide to participate, you will join a study funded by the National Institute of Health and you will be assigned to one of the ASU SIBS afterschool programs. These programs are focused on working with sisters and brothers to learn and practice new skills and participate in educational activities. In each group, your children will participate in a series of 12 group meetings as an afterschool program, each lasting 90 minutes and including hands-on group activities, games, and discussions. Your family will also be invited to three Family Fun nights, where we will show you what your children have been learning in the afterschool sessions.

Regardless of which group you are assigned to, you and your children will be asked to participate in three interviews, once before the program begins, a second interview after the program ends, and a third interview 12 months later. These interviews will take place over the phone for parents and in the afterschool setting or in the home for children. Each will last about 60 minutes and ask about you and your children's behaviors, feelings, relationships, and school experiences. In addition, your children will be asked to participate in 7 nightly phone calls, each lasting about 10 minutes to find out about their daily activities and feelings, before the program and after the program ends. You will be contacted by the Pennsylvania State University Survey Research Center for these phone calls. At the final family night, we will ask you to complete an anonymous survey about your experiences in the program, which takes about five minutes.

#### **VIDEO RECORDING AND PHOTOGRAPHS OF STUDY ACTIVITIES**

The research team will videotape and photograph study activities to assist with researcher training, evaluate research activities, and for use in research presentations. All video files will be stored indefinitely on a password-protected computer server.

#### RELEASE OF SCHOOL RECORDS AND PERMISSION TO CONTACT TEACHERS

The research team is requesting your permission to release your children's school records exclusively for research purposes. This information will be used to examine if the intervention is having positive effects on your children's school adjustment. As with all study data, this information will be maintained confidential and your children's names will never be disclosed in research reports. In addition, the research team is requesting your permission to contact your children's teachers in order to request their evaluations of your children.

#### RISKS

This study involves minimal risk; that is, no risks to your physical or mental health beyond those encountered in the normal course of everyday life. There are personal questions in the surveys which may cause discomfort for some individuals.

| В | E | N | Е | F | Π | S |
|---|---|---|---|---|---|---|

| Family ID: |
|------------|

Benefits of this program may include warmer and closer sibling and family relationships. The development of this program may also benefit future participants. No benefit to you from this research can be guaranteed.

#### CONFIDENTIALITY

All information obtained in this study is strictly confidential. The results of this research study may be used in reports, presentations, and publications, but the researchers will not identify you or your child. In order to maintain confidentiality of your records, Dr. Updegraff will use the following procedures: all data collected will be labeled with numerical codes and your names will not be attached to this information. The key to the code will be kept in a locked drawer and only members of the research team will have access to it. You further understand that all data is kept indefinitely and used for research only.

In order to keep your answers private, we also have a Certificate of Confidentiality from the U.S. Government. which protects us from having to share any information that may identify you, or any of the information you give us, even if it is requested for federal, state, or local civil, criminal or other proceedings.

You understand that all the information obtained in this study will be kept confidential with two exceptions:

- a. You understand that if, during the interview, there is evidence of extreme depression or potential suicide, the Project staff will work with you and a local agency to see that either of you or your children get the help you (or they) need. In this case, one of the project staff would talk with professionals at the mental health agency who would then contact you about getting help.
- b. You also understand that the project staff is required by law to report to appropriate authorities any report of child abuse of your minor children.

A description of this project will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### WITHDRAWAL PRIVILEGE

Participation in this study is completely voluntary. It is ok for you to say no. Even if you say yes now, you are free to say no later, and withdraw from the study at any time. Your decision will not affect your relationship with Arizona State University or your child's school.

### **COSTS AND PAYMENTS**

You will receive \$20 for the home visit today, and each participating parent will receive \$35 for the first interview, \$40 for the second interview, and \$50 for the third interview. Parents will receive an additional \$35 (beginning of study) and \$40 (after the program) for their children's participation in the 7 phone calls.

#### **VOLUNTARY CONSENT**

Please carefully read the following four statements, indicate your response, and initial in the space

| provided: | mig four statements, ma | iodic your response, and initial in the space |
|---|---|---|
| I consent to video recording of my | children and my family for r | esearch purposes as described above: |
| Yes | No | _ (initials here) |
| I consent to photographs of my ch | ldren and my family for rese | earch purposes as described above: |
| Yes | No | _ (initials here) |
| I consent to the release of both of to be used exclusively for research | | s to the research team, led by Dr. Kim Updegraff, |

Family ID:

| | Yes | No | (initials here) | |
|---|---|---|---|---|
| I give permiss | sion to the research tea | m, led by Dr. Kim Updegra | aff, to contact my chi | ildren's teachers: |
| | Yes | No | (initials here) | |
| are satisfied y<br>happy to answ<br>contact Dr. Ki | ou understand this forr<br>wer any questions you h | | its risks and benefit<br>If you have any ques | |
| placed at risk | ; you can contact the C | nts as a subject/participant<br>hair of the Human Subject<br>urance, at 480-965 6788. | | if you feel you have been<br>w Board, through the ASU |
| knowingly to a participate or benefit. In sign | assume any risks involv<br>to withdraw your conse | • | icipation is voluntary<br>pation at any time wi | y. You may choose not to |
| • | e indicates that you cor<br>the above study. | nsent for you and your chil | dren (5 <sup>th</sup> grader, you | unger sister or brother) to |
| Name of Parti | icipating 5 <sup>th</sup> Grader (Ple | ease print) | | |
| Name of Parti | icipating Younger Siste | r or Brother (Please print) | | |
| Name of Pare | ent/Legal Guardian (Ple | ase print) | | |
| Name of Seco | ond Parent/Legal Guard | dian – if participating (Plea | se print) | |
| Signature of F | Parent/Legal Guardian | | | <br>Date |
| Signature of S | Second Parent/Legal G | uardian – if participating | | <br>Date |
| "I certify that I<br>possible risks<br>been raised, a<br>Assurance giv | associated with partici<br>and have witnessed the<br>ven by Arizona State Ui | | dy, have answered a<br>elements of Informed<br>uman Research Pro | any questions that have |
| Signature of I | nvestigator | | Date | |
| | | | Family ID | : |

# ASU SIBS Project Arizona State University T. Denny Sanford School of Social and Family Dynamics

Hoja de Consentimiento Informado para Padres/Tutores y Menores de Edad

#### INTRODUCCIÓN

El propósito de esta forma es para proporcionarle a usted (como un futuro participante) información que podría afectar su decisión de participar o no en esta investigación, y para registrar el consentimiento de aquellas personas que aceptan estar involucradas en el estudio.

#### **INVESTIGADORA**

La Doctora Kimberly Updegraff, profesora de la Facultad de Desarrollo Humano y de la Familia en la Universidad Estatal de Arizona (ASU), le ha invitado a usted a participar en un estudio de investigación.

# DESCRIPCIÓN DEL ESTUDIO DE INVESTIGACIÓN

El propósito de la investigación es evaluar la efectividad de un programa que promueva relaciones positivas entre hermanos(as) y entre la familia, entre compañeros(as), y la adaptación escolar. Si usted decide participar, se unirá a una investigación patrocinada por el Instituto Nacional de Salud, y usted será asignado a uno de los programas de ASU SIBS que se llevará a cabo después de la escuela. Estos programas se enfocan en trabajar con hermanas y hermanos para aprender y practicar nuevas habilidades y participar en actividades educativas. En cada grupo, sus hijos participarán en una serie de 12 reuniones grupales como parte de un programa después de clases, cada reunión dura 90 minutos e incluye actividades grupales interactivas, juegos, y pláticas. Su familia también será invitada a tres Noches de Diversión para las Familias donde les enseñaremos lo que sus hijos(as) han estado aprendiendo en las sesiones después de clases.

Independientemente del grupo al que usted sea asignado(a), se les va a pedir a usted y a sus hijos que participen en tres entrevistas, una vez antes de que el programa comience, una segunda entrevista después de que finalice el programa y una tercera entrevista 12 meses después. Estas entrevistas serán por teléfono para los padres, y en la escuela después de clases o en las casas para los niños. Cada entrevista durará aproximadamente 60 minutos y se le preguntará sobre usted y sobre los comportamientos de sus hijos(as), sus sentimientos, relaciones, y experiencias escolares. También, se les pedirá a sus hijos que participen en 7 llamadas telefónicas cada noche, de 10 minutos cada una, para conocer sobre sus actividades diarias y sus sentimientos, antes del programa y después de que finalice el programa. El Centro de Investigación de Encuestas de la Universidad Estatal de Pensilvania se comunicará con usted sobre estas llamadas telefónicas. En la última noche de diversión para las familias, le pediremos que complete una encuesta anónima acerca de sus experiencias en el programa la cual tomará unos cinco minutos.

# GRABACIÓN EN VIDEO Y FOTOGRAFIAS DE LAS ACTIVIDADES DEL ESTUDIO

El equipo de investigación grabará en video y con fotografía las actividades del estudio para ayudar con la formación de los investigadores, para evaluar las actividades de la investigación,

| Famil | lv ID: |
|-------|--------|

y para el uso en las presentaciones de la investigación. Todos los archivos de vídeo serán guardados indefinidamente en un servidor de computadora protegido con una contraseña.

# <u>OBTENCIÓN DE LOS REGISTROS ESCOLARES Y PERMISO PARA COMUNICARNOS</u> CON LOS MAESTROS

El equipo de investigación está solicitando su permiso para obtener los registros escolares de sus hijos exclusivamente para los fines de la investigación. Esta información será usada para examinar si la intervención está teniendo efectos positivos en la adaptación escolar de sus hijos. Al igual que con todos los datos del estudio, esta información se mantendrá confidencial y los nombres de sus hijos nunca se divulgarán en los informes de investigación. El equipo de investigación también está solicitando su permiso para comunicarse con los maestros de sus hijos para solicitar las evaluaciones de sus hijos.

#### **RIESGOS**

Este estudio tiene riesgos mínimos; esto significa que no hay riesgos para su salud física o mental más allá de los que se encuentran en el curso normal de la vida diaria. Sin embargo, hay preguntas personales en las encuestas que le podrían causar incomodidad a algunos individuos.

#### **BENEFICIOS**

Algunos beneficios de este programa podrían incluir relaciones más cálidas entre hermanos(as) y familiares. El desarrollo de esta investigación también podrá beneficiar a futuros participantes. No se puede garantizar ningún beneficio para usted de esta investigación.

### **CONFIDENCIALIDAD**

Toda la información obtenida en este estudio es estrictamente confidencial. Los resultados de esta investigación podrán ser usados en reportes, presentaciones, y publicaciones, pero los investigadores no los identificará ni a usted ni a sus hijos. Para mantener la confidencialidad de su información, la Dra. Updegraff hará lo siguiente: marcará todos los datos recopilados con un código numérico y sus nombres no serán puestos junto a este código. La clave para el código estará guardada en un cajón cerrado con llave y solamente los miembros del equipo de investigación tendrán acceso a la misma. Adicionalmente, usted entiende que todos los datos serán guardados indefinidamente y usados solamente para propósitos de la investigación.

Para mantener sus respuestas privadas, además tenemos un Certificado de Confidencialidad del Gobierno de Estados Unidos que nos protege a nosotros de tener que compartir cualquier tipo de información que pueda identificarlo(a) a usted o a la información que nos ha dado, aún si la misma es solicitada para algún procedimiento federal, estatal, o local civil, penal, o de otro tipo.

Usted entiende que toda la información que se obtenga en este estudio se mantendrá confidencial con solo dos excepciones:

a. Usted entiende que si, durante la entrevista, hay evidencia de depresión severa o suicidio potencial, el personal del Proyecto trabajará con usted y con una agencia local para encontrarles a ustedes o a sus hijos la ayuda que ustedes (o ellos) necesiten. Uno de los miembros del equipo del proyecto hablará con los profesionales en la agencia de salud mental, quienes luego se pondrán en contacto con usted para

| Family | ID· |
|--------|-----|
| ганні | 111 |

proporcionales ayuda.

b. Usted también entiende, que por ley, se le exige al personal del proyecto que reporte a las autoridades apropiadas si hay algún caso de abuso de niños menores de edad.

Una descripción de este proyecto estará disponible en la página de internet: http://www.ClinicalTrials.gov, tal como lo exige la ley de EE. UU. Esta página de internet no incluirá información que pueda identificarlos. Como máximo, la página de internet incluirá un resumen de los resultados. Usted puede mirar esta página de internet en cualquier momento.

#### PRIVILEGIO DE RETIRARSE

La participación en este estudio es completamente voluntaria. Está bien que usted diga no. Aunque usted diga que sí ahora, está libre de decir no más tarde, y retirarse del estudio en cualquier momento. Su decisión no afectará su relación con ASU ni con la escuela de sus hijos(as).

# **COSTO Y PAGOS**

Usted recibirá \$20 por la visita de hoy a su casa y cada padre participante recibirá \$35 por la primera entrevista, \$40 por la segunda entrevista y \$50 por la tercera entrevista. Los padres recibirán \$35 adicionales (al comienzo del estudio) y \$40 (después del programa) por la participación de sus hijos en las 7 llamadas telefónicas.

### **CONSENTIMIENTO VOLUNTARIO**

Por favor, lea atentamente las siguientes cuatro declaraciones, indique su respuesta y escriba sus iniciales en el espacio provisto:

| • | sentimiento a la grabació<br>on como se describe ante | ón de video de mis hijos y mi familia co<br>eriormente: | on fines de |
|---|---|---|---|
| Sí | No | (iniciales aquí) | |
| • | sentimiento a las fotogra | fías de mis hijos y mi familia con fines | de investigación |
| Sí | No | (iniciales aquí) | |
| equipo de in | | registros escolares de mis dos hijos(a<br>la Dra. Kim Updegraff, para que sean<br>investigación: | |
| Sí | No | (iniciales aquí) | |
| Doy permis<br>maestros de | | ción, dirigido por la Dra. Kim Updegrafi | f, para contactar a los |
| Sí | No | (iniciales aquí) | |
| y (b) que us | sted está satisfecho(a) de | iendo: (a) que ha leído esta forma o se<br>e que comprende esta forma, el estudi<br>igadores estarán disponibles para resp | io de investigación y |
| | | | Family ID: |

pregunta que usted tenga sobre la investigación. Si tiene alguna pregunta, no dude en ponerse en contacto con la Dra. Kimberly Updegraff. Ella puede ser contactada por teléfono al 480-965-6669, o por correo electrónico a Kimberly.updegraff@asu.edu.

Si usted tiene alguna pregunta sobre sus derechos como sujeto/participante en esta investigación, o si siente que lo han puesto en riesgo, puede comunicarse con el presidente de la Junta Institucional de Revisión de los Sujetos Humanos, a través de la Oficina de Protección e Integridad de la Investigación de ASU al (480) 965-6788.

Esta forma explica la naturaleza, el propósito, los beneficios y todos los riesgos asociados con el proyecto. Al firmar esta forma, usted está de acuerdo que asume cualquier riesgo asociado con su participación. Recuerde, su participación es voluntaria. Usted puede elegir no participar o retirarse en cualquier momento sin ninguna penalidad y sin pérdida de beneficios. Al firmar esta forma de consentimiento, usted no está renunciando sus derechos legales. Se le dará (ofrecerá) una copia firmada de esta forma de consentimiento.

Su firma indica su consentimiento para que usted y sus hijos(as) (un(a) estudiante en el 5º

grado, y un(a) hermano(a) menor) participen en el estudio mencionado arriba. Nombre del/de la participante de 5° grado (Por favor escriba en letra molde) Nombre del hermano(a) menor que participa (Por favor escriba en letra molde) Nombre del padre/madre/tutor legal (Por favor escriba en letra molde) Nombre del padre/madre/tutor legal – Si participa (Por favor escriba en letra molde) Firma del padre/madre/tutor legal Fecha Firma del padre/madre/tutor legal - Si participa Fecha **DECLARACIÓN DE LA INVESTIGADORA** "Certifico que este estudio de investigación ha sido explicado a la persona arriba mencionada por mi personal de investigación. La persona entiende la naturaleza y el propósito, y los posibles riesgos y beneficios asociados con esta investigación. Cualquier pregunta ha sido respondida y la entrevistadora ha atestiguado dicha firma. Estos elementos del acuerdo informado se conforman a la garantía dada por la Universidad Estatal de Arizona (ASU) al Departamento de Salud y Servicios Humanos (DHHS) para proteger los derechos de sujetos humanos. Le he proporcionado (ofrecido) al sujeto/participante una copia de este documento de consentimiento firmado." Firma de la Investigadora Fecha Family ID:

Child Assent - 5th Grader

I have been told that my parent/legal guardian has said it is okay for me to take part in this project about families and activities.

I will participate in an afterschool program with my younger sister or brother. The afterschool program will take place one day a week at my school for 12 weeks, and each session will last about 90 minutes. My family will also be invited to attend three family nights so that my parents can learn about what I am doing in the afterschool program. I will be asked to participate in three interviews during a 90-minute afterschool session. I will do the first interview at the beginning of the project, the second interview at the end of the project, and the third interview will be done about 12 months after the program ends. I will also be asked to participate in 7 nightly phone calls, lasting about 10 minutes each, before the program begins and after the program ends. Someone from Pennsylvania State University will call me for these phone calls.

I am taking part in this program because I want to. I know that I can stop at any time if I want to and it will be okay if I want to stop.

| Print Your Name | |
|-----------------|---|
| Sign Your Name | |
| Date | _ |
| Date | |

| 1 | | • 1 | T1 | |
|---|------|-----|------|-----|
| ı | Fam | 111 | 7 | ١. |
| ı | rann | 11 | v ii | IJ. |

Hoja de Asentimiento - Estudiante de 5º grado

Me han dicho que mi madre/padre/tutor dijo que está bien que yo tome parte en este proyecto sobre familias y actividades.

Participaré en un programa después de la escuela con mi hermano o hermana menor. El programa después de la escuela se llevará a cabo un día a la semana en mi escuela durante 12 semanas, y cada sesión durará aproximadamente 90 minutos. Mi familia también será invitada a asistir a tres noches familiares para que mis padres se puedan enterar de lo que estoy haciendo en el programa después de la escuela. Se me pedirá que participe en tres entrevistas durante una sesión extracurricular de 90 minutos. Haré la primera entrevista al comienzo del proyecto, la segunda entrevista al final del proyecto, y la tercera entrevista se realizará aproximadamente 12 meses después de que finalice el programa.

Estoy participando en este programa porque quiero. Yo sé que puedo parar en cualquier momento, si quiero, y que estará bien si decido parar.

| laniny ID. | Famil | / ID: |
|------------|-------|-------|
|------------|-------|-------|

Child Assent - Younger Sister/Brother

I have been told that my parent/legal guardian has said it is okay for me to take part in this project about families and activities.

I will participate in an afterschool program with my older sister or brother. The afterschool program will take place one day a week at my school for 12 weeks, and each session will last about 90 minutes. My family will also be invited to attend three family nights so that my parents can learn about what I am doing in the afterschool program. I will be asked to participate in three interviews during a 90-minute afterschool session. I will do the first interview at the beginning of the project, the second interview at the end of the project, and the third interview will be done about 12 months after the program ends. I will also be asked to participate in 7 nightly phone calls, lasting about 10 minutes each, before the program begins and after the program ends. Someone from Pennsylvania State University will call me for these phone calls.

I am taking part in this program because I want to. I know that I can stop at any time if I want to and it

| will be okay if I want to stop. | • |
|---------------------------------|---|
| Print Your Name | |
| Sign Your Name | |
| Date | |

| Famil | ly I | D: |
|-------|------|----|

Hoja de Asentimiento – Hermano/a Menor

Me han dicho que mi madre/padre/tutor dijo que está bien que yo tome parte en este proyecto sobre familias y actividades.

Participaré en un programa después de la escuela con mi hermano o hermana menor. El programa después de la escuela se llevará a cabo un día a la semana en mi escuela durante 12 semanas, y cada sesión durará aproximadamente 90 minutos. Mi familia también será invitada a asistir a tres noches familiares para que mis padres se puedan enterar de lo que estoy haciendo en el programa después de la escuela. Se me pedirá que participe en tres entrevistas durante una sesión extracurricular de 90 minutos. Haré la primera entrevista al comienzo del proyecto, la segunda entrevista al final del proyecto, y la tercera entrevista se realizará aproximadamente 12 meses después de que finalice el programa.

Estoy participando en este programa porque quiero. Yo sé que puedo parar en cualquier momento, si quiero, y que estará bien si decido parar.

| Escribe tu nombre |
|-------------------|
| Firma tu nombre |
| Fecha |

| Famil <sup>1</sup> | v ID. |
|--------------------|-------|